CLINICAL TRIAL: NCT00969774
Title: Facial Type Determination Through Ricketts Cephalometric Analysis, Anthropometric Measurements, Indices and Proportions and Facial Analysis Performed by Means of Photographs
Brief Title: Facial Type Determination Through Cephalometry, Anthropometry and Facial Analysis
Status: Completed | Type: Observational
Sponsor: Pontificia Universidade Catolica de Sao Paulo (Other)
Responsible Party: Rossana Ribeiro Ramires, Pontificia Universidade Catolica de Sao Paulo
Other Study IDs: PUC/SP 0021/2006
Record Dates: First submitted 2009-08-31; First posted 2009-09-01 (Estimated); Last update posted 2009-09-02 (Estimated); Status verified 2009-09

CONDITIONS: Healthy
Keywords: Face; Cephalometry; Anthropometry; Photography; Diagnosis; Adult; Morphology; Comparative Study
MeSH Terms: conditions — Facies; Disease

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Cross-Sectional
Oversight: Data Monitoring Committee: Yes

SUMMARY:
Introduction:

Human face with its bony and muscular structures has singular and peculiar characteristics. It may be classified in three types, associated with the variation of shape and craniofacial configuration, both in vertical and horizontal planes, directly affecting dental occlusion, face harmony, orofacial musculature and oral functions. Aim: to correlate cephalometric with anthropometric and facial analysis findings on determining the facial type.

Method:

105 leukoderm adults were involved, 34 male and 71 female aging between 20 and 40 years old. Data were collected in December 2006 in an orthodontic clinic located at Belo Horizonte- MG, Brazil. Cephalometric findings to determinate facial types were compared to seven anthropometric facial measurements, three anthropometric facial proportions and three anthropometric facial indices, in addition to facial type identification through clinical facial analysis of photographs.

ELIGIBILITY:
Inclusion Criteria:

* to have Ricketts cephalometric analysis

Exclusion Criteria:

* to have been submitted on orthognathic surgery
* black or asian people

Ages: 20 Years to 40 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Study Population: primary care orthodontic clinic
Sampling Method: Probability Sample
Enrollment: 105 (Actual)
Dates: Start 2006-02; Primary Completion 2006-11 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Rossana R Ramires, MSc, Principal Investigator — Pontifícia Universidade Católica de São Paulo